CLINICAL TRIAL: NCT04739891
Title: Acute Cholecystitis With Concomitant Choledocholithiasis: Unicentric Study of Prevalence and Predictive Factors for Its Diagnosis and Management
Brief Title: Acute Cholecystitis With Concomitant Choledocholithiasis: Unicentric Study of Prevalence and Predictive Factors
Acronym: CHOLEPREV
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospital de Mataró (Other)
Responsible Party: Principal Investigator, Ana Ciscar, General and digestive surgery specialist, Hospital de Mataró
Other Study IDs: CHOLEPREV2021
Record Dates: First submitted 2021-02-01; First posted 2021-02-05 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Acute Cholecystitis; Choledocholithiasis
Keywords: Acute Cholecystitis; Choledocholithiasis; Urgent cholecystectomy; Risk factors
MeSH Terms: conditions — Cholecystitis, Acute; Choledocholithiasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The management of cholelithiasis with choledocolithiasis is extensively known, whereas for Acute Calculous Cholecystitis (ACC) with choledocolithiasis or common bile duct stones (CBDS), a common entity, there is a lack of protocols for optimising treatment. The main hypothesis of our study is: a correct stratification of the concomitant CBDS probability at ACC diagnosis would optimize its treatment as early targeted treatment could be performed. One-step management of ACC with CBDS by a specialised hepatobiliary team would represent a benefit to the patient in terms of morbi-mortality, admission time and number of admissions. The aim of our study is to identify high / intermediate probability criteria for CBDS associated when diagnosing CA. This is a retrospective study of patients who were operated on with an emergent cholecystectomy in our center from 01/2012 to 12/2019.

DETAILED DESCRIPTION:
Data will be obtained from the hospital (Consorci Sanitari del Maresme) clinical database.

The Ethics Committee approval has been obtained.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years

Exclusion Criteria:

* Non urgent cholecystectomy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients who underwent emergent cholecystectomy for acute calculous cholecystitis
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-02-15 (Estimated); Primary Completion 2021-04-15 (Estimated); Study Completion 2021-04-15 (Estimated)

PRIMARY OUTCOMES:
CBDS risk | From diagnostic to surgery
  Probability of CBDS presence at the moment of AC diagnose based on classification on risk modified from Maple et al. 2010: high, intermediate or low

SECONDARY OUTCOMES:
Intraoperative cholangiography | During the surgery
  Percentage of patients who underwent intraoperative cholangiography (IOC) in each group: %
Postoperative morbidity | From surgery to 1 year
  Adverse events (biliary fistula presence and ERCP (endoscopic retrograde cholangiopancreatography) requirements) identification during the postoperative period: Y/N
Readmission | From discharge to 1 year
  Requirement of readmission after discharge

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pisano M, Allievi N, Gurusamy K, Borzellino G, Cimbanassi S, Boerna D, Coccolini F, Tufo A, Di Martino M, Leung J, Sartelli M, Ceresoli M, Maier RV, Poiasina E, De Angelis N, Magnone S, Fugazzola P, Paolillo C, Coimbra R, Di Saverio S, De Simone B, Weber DG, Sakakushev BE, Lucianetti A, Kirkpatrick AW, Fraga GP, Wani I, Biffl WL, Chiara O, Abu-Zidan F, Moore EE, Leppaniemi A, Kluger Y, Catena F, Ansaloni L. 2020 World Society of Emergency Surgery updated guidelines for the diagnosis and treatment of acute calculus cholecystitis. World J Emerg Surg. 2020 Nov 5;15(1):61. doi: 10.1186/s13017-020-00336-x. PMID 33153472